CLINICAL TRIAL: NCT00747903
Title: Investigation of the Effectiveness of Non-Coherent Blue Light in Intralesional Photodynamic of Basal Cell Carcinoma
Brief Title: Photodynamic Therapy Using Aminolevulinic Acid in Treating Patients With Skin Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laser and Skin Surgery Center of New York (Other)
Responsible Party: Roy G. Geronemus, Laser and Skin Surgery Center of New York
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000613601; DUSA-PDT-BCC-06
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-07

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; recurrent skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — Aminolevulinic Acid

INTERVENTIONS:
Drug: aminolevulinic acid hydrochloride

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. This may be an effective treatment against skin cancer.

PURPOSE: This phase II trial is studying the side effects of photodynamic therapy using aminolevulinic acid and to see how well it works in treating patients with skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the safety and efficacy of intralesional photodynamic therapy using aminolevulinic acid and non-coherent blue light in patients with nodular basal cell carcinoma.

OUTLINE: Patients undergo photodynamic therapy comprising intralesional injection of aminolevulinic acid followed by non-coherent blue light therapy over approximately 17 minutes. Patients may undergo re-treatment with photodynamic therapy 8 weeks later.

Patients undergo photographic assessment of their skin lesions at baseline, 8 weeks, 16 weeks, and then at 1 and 2 years to evaluate healing time, clinical improvement, and side effects.

Patients undergo biopsies of their skin lesions at 16 weeks and then at 1 and 2 years to confirm histological clearance.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven basal cell carcinoma on the trunk or extremities

  * Tumor size ≤ 2 cm in diameter

PATIENT CHARACTERISTICS:

* Willing and able to comply with all follow-up requirements
* Mentally competent
* No active, localized, or systemic infections
* Not immunocompromised
* No coagulation disorder
* No photosensitivity or allergy to sunlight
* Not pregnant or nursing
* No history of keloid formation
* No history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins, or photodermatosis

PRIOR CONCURRENT THERAPY:

* No prior gold therapy
* No prior radiotherapy to the trunk and extremities
* More than 24 months since prior oral retinoids (e.g., isotretinoin or acitretin) or photosensitizing drugs (e.g., Declomycin®)
* More than 1 year since prior collagen or other injections, Botox® injections, chemical peels, dermabrasion, or resurfacing procedures
* More than 1 month since prior topical retinoid therapy
* No concurrent aspirin or antioxidants
* No concurrent anticoagulation medications

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Diana Santanello — Laser and Skin Surgery Center of New York
Locations (1):
- Laser and Skin Surgery Center of New York, New York, New York, United States